CLINICAL TRIAL: NCT00012870
Title: Effect of Behavioral Management on Quality of Life in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: NRI 95-244
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Behavioral Management

INTERVENTIONS:
Behavioral: Behavioral Management

SUMMARY:
Nurses play an important role in helping patients to manage symptoms, adhere to treatment, and change behavior. There has been a lack of research regarding nonpharmacologic interventions with patients with heart failure and other chronic conditions.

DETAILED DESCRIPTION:
Background:

Nurses play an important role in helping patients to manage symptoms, adhere to treatment, and change behavior. There has been a lack of research regarding nonpharmacologic interventions with patients with heart failure and other chronic conditions.

Objectives:

The primary objective of this 4-year study was to determine the effect of a nurse-led behavioral management intervention on health-related quality in patients with medically-managed heart failure. The secondary objective was to assess the impact of the behavioral management intervention on health care resource utilization.

Methods:

DESIGN: randomized controlled trial. SETTING: single site, VA San Diego Healthcare System. SAMPLE: Patients were enrolled in 11 cohorts a total of 116 outpatients were randomly assigned to one of two treatment groups to evaluate the clinical impact of the intervention. Group 1 received usual care for patients with heart failure (n=58). Group 2 was an augmented group receiving usual care plus participation in the 15-week (4-month) behavioral management program (n=58). Inclusion criteria were that the patient had a primary diagnosis of heart failure, a VA primary care provider, stable symptoms for at least one month and was able to walk. INTERVENTION: The behavioral management program augmented usual care and consisted of establishing specific goals with patients related to healthier diet, increased quality and amount of exercise, smoking cessation, and increased social and interpersonal activities. DEPENDENT VARIABLES/OUTCOME MEASURES: The five major dependent variables for this study were psychological symptom distress (Multiple Affect Adjective Check List - MAACL), physical functioning (SF-36 physical component summary score), mental functioning (SF-36 mental component summary score), exercise capability (6-Minute Walk), and general health perceptions (SF-36 general health scale score). Dependent variables were assessed at baseline, at the end of treatment (at 4 months), and then at 10 and 16 months. DATA ANALYSIS: Initial analyses included all subjects who were randomized to treatment and completed all data collection time points in a series of 2 by 4 ANOVAs with time as a repeated measure.

Status:

Completed. Final report submitted August 2003

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are that the patient has a primary diagnosis of dilated cardiomyopathy or heart failure, a VA primary care provider, stable symptoms for at least one month and is able to walk.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha J. Shively, PhD RN, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Result] Shively M, Kodiath M, Smith TL, Kelly A, Bone P, Fetterly L, Gardetto N, Shabetai R, Bozzette S, Dracup K. Effect of behavioral management on quality of life in mild heart failure: a randomized controlled trial. Patient Educ Couns. 2005 Jul;58(1):27-34. doi: 10.1016/j.pec.2004.06.007. PMID 15950833
- [Result] Shively M, Fox C, Brass-Mynderse NJ. Health-related quality of life as an outcome for patients with heart failure. J Cardiovasc Nurs. 1996 Jan;10(2):89-96. doi: 10.1097/00005082-199601000-00009. PMID 8656241
- [Result] Kodiath M, Kelly A, Shively M. Improving quality of life in patients with heart failure: an innovative behavioral intervention. J Cardiovasc Nurs. 2005 Jan-Feb;20(1):43-8. doi: 10.1097/00005082-200501000-00009. PMID 15632812